CLINICAL TRIAL: NCT00238173
Title: Phase I Dose Escalation Study of N-Acetylcysteine Administered in Conjunction With Carboplatin, Cyclophosphamide, and Etoposide Phosphate BBBD, in Children With Malignant Brain Tumors
Brief Title: Acetylcysteine, Mannitol, Combination Chemotherapy, and Sodium Thiosulfate in Treating Children With Malignant Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: OHSU IRB closed study to further enrollment 2/17/2006
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002050; OHSU-8522; OHSU-SOL-04085-L; OHSU-IRB-2050
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Bone Marrow Suppression; Brain and Central Nervous System Tumors; Drug/Agent Toxicity by Tissue/Organ; Long-term Effects Secondary to Cancer Therapy in Children
Keywords: drug/agent toxicity by tissue/organ; bone marrow suppression; long-term effects secondary to cancer therapy in children; recurrent childhood brain stem glioma; untreated childhood brain stem glioma; childhood central nervous system germ cell tumor; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood brain tumor; recurrent childhood cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; childhood oligodendroglioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood ependymoma; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor; recurrent childhood central nervous system embryonal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Drug-Related Side Effects and Adverse Reactions; Optic Nerve Glioma; Astrocytoma; Medulloblastoma; Oligodendroglioma; Familial ependymoma | interventions — Filgrastim; Acetylcysteine; Carboplatin; Cyclophosphamide; etoposide phosphate; Mannitol; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: acetylcysteine — administered i.v. over 30 to 60 minutes
Drug: carboplatin — (200 mg/m2/day; total dose 400 mg/m2) will be infused i.a. over 10 minutes, in 50-180 cc of normal saline.
Drug: cyclophosphamide — (330 mg/m2/day; total dose 660 mg/m2) will be infused i.v. in 25-50 cc of normal saline, over approximately 10 minutes.
Drug: etoposide phosphate — (200 mg/m2/day; total dose 400 mg/m2) will be infused i.v. in 25-100 cc of normal saline, over approximately 10 minutes, immediately following the cyclophosphamide.
Drug: mannitol — (25%) delivered i.a. at a pre-determined flow rate over 30 seconds. The flow rate will be determined by iodinated contrast injection and fluoroscopy as the lowest infusion rate in which there is retrograde flow from the arterial catheter. The rate and volume of mannitol infused will be approximately 4-12 cc/sec x 30 seconds.
Drug: sodium thiosulfate — STS is available as a 25% (250 mg/ml) solution. The dose of STS administered 4 hours after carboplatin is 16 gm/m2. The dose of STS administered 8 hours after carboplatin is 16 gm/m2. Actual dose to be administered will be determined and mixed with an equivalent amount of sterile water (1 ml:1 ml) for infusion.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, etoposide phosphate, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Mannitol may help chemotherapy work better by making it easier for these drugs to get to the tumor. Chemoprotective drugs, such as acetylcysteine and sodium thiosulfate, may protect normal cells from the side effects of chemotherapy. Giving acetylcysteine together with mannitol, combination chemotherapy, and sodium thiosulfate may be an effective treatment for malignant brain tumors.

PURPOSE: This phase I trial is studying the side effects and best dose of acetylcysteine when given together with mannitol, combination chemotherapy, and sodium thiosulfate in treating children with malignant brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity and maximum tolerated dose of acetylcysteine when given in combination with blood-brain barrier disruption treatment with mannitol, combination chemotherapy comprising cyclophosphamide, etoposide phosphate, and carboplatin, and delayed high-dose sodium thiosulfate in pediatric patients with malignant brain tumors.

Secondary

* Determine the blood/bone marrow toxicity of this regimen in these patients.
* Determine tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of acetylcysteine.

Patients receive acetylcysteine IV over 30-60 minutes followed, at least 15 minutes later, by x-ray-guided femoral artery catheterization under general anesthesia on days 1 and 2. After placement of the catheter, patients receive cyclophosphamide IV over 10 minutes, etoposide phosphate IV over 10 minutes, mannitol intra-arterially (IA) over 30 seconds, and carboplatin IA over 10 minutes also on days 1 and 2. Patients then receive high-dose sodium thiosulfate IV over 15 minutes 4 hours after completion of carboplatin. Some patients may receive a second dose of sodium thiosulfate 8 hours after completion of carboplatin. Beginning 48 hours after the last dose of chemotherapy on day 2, patients receive filgrastim (G-CSF) subcutaneously once daily for 7-10 days or until blood counts recover. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of acetylcysteine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 3 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed brain tumors, including any of the following:

  * Brain stem glioma
  * Primitive neuroectodermal tumor
  * CNS germ cell tumor
  * Malignant glioma
* Diagnosis based on any of the following:

  * CT-assisted or stereotactic biopsy
  * Open biopsy
  * Surgical resection
  * Cerebrospinal fluid cytology
  * Elevated tumor markers
  * Unequivocal radiographic changes (for patients with brain stem glioma or optic glioma)
* All tumor types, except brain stem glioma, must be recurrent
* No radiographic signs of intracranial herniation and/or spinal cord block

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 90 days

Hematopoietic

* WBC ≥ 2,500/mm^3
* Absolute granulocyte count ≥ 1,200/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT and SGPT < 2.5 times upper limit of normal
* Bilirubin < 2.0 mg/dL

Renal

* Creatinine < 1.8 mg/dL

Pulmonary

* No history of clinically significant reactive airway disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant risk for general anesthesia
* No uncontrolled, clinically significant, confounding medical condition within the past 30 days
* No contraindication to study drugs

PRIOR CONCURRENT THERAPY:

Chemotherapy

* At least 28 days since prior systemic chemotherapy

Radiotherapy

* At least 3 months since prior total spine radiotherapy
* At least 14 days since prior cranial radiotherapy
* Prior systemic radiotherapy allowed

Surgery

* See Disease Characteristics

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2004-12; Primary Completion 2006-02-17 (Actual); Study Completion 2006-02-17 (Actual)

PRIMARY OUTCOMES:
To assess toxicity and the maximally tolerated dose of N-acetylcysteine administered in conjunction with carboplatin, cyclophosphamide and etoposide phosphate BBBD, and delayed high dose sodium thiosulfate, in children with malignant brain tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States